CLINICAL TRIAL: NCT01883453
Title: A Double Blinded Clinical Study Aiming to Shorten an Episode of Common Cold When the Treatment is Started at the Onset of an Episode of Common Cold
Brief Title: A Nasal Spray With Glucose Oxidase as a Treatment of Common Cold
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Krister Tano, MD, PhD, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GOcoldU&B2013
Record Dates: First submitted 2013-04-23; First posted 2013-06-21 (Estimated); Results first posted 2015-11-09 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-06

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline+glucose nasal spray (Placebo Comparator): A nasal spray with isotone saline + 5% glucose, dosing one puff 5 times daily in each nostril at the first treatment day and thereafter trice daily for a total of one week
  Interventions: Device: Saline+5%glucose
- Nasal spray with glucose oxidase+glucose (Active Comparator): A nasal spray with 200U/ml of glucose oxidase + 5% glucose. Treatment starts with 5 puffs in each nostril at the first day, and thereafter trhee times daily for a total treatment time of one week.
  Interventions: Device: Glucose oxidase+5%glucose

INTERVENTIONS:
Device: Glucose oxidase+5%glucose — A hydrogen peroxide producing enzyme
  Arms: Nasal spray with glucose oxidase+glucose
Device: Saline+5%glucose — Isotonic saline + 5% glucose in a bag-on-valve nasal spray device
  Arms: Saline+glucose nasal spray

SUMMARY:
Healthy persons are invited to participate in the study and are given a home protocol (WURSS21), nasal spray and a sample pin. The included persons are told to make a nasopharyngeal sampling from the nose when they are sure that they have caught a common cold. After the sampling they start to spray and also fill in the records daily. The aim of the study is to investigate whether a nasal spray with glucose oxidase could shorten an episode of common cold.

DETAILED DESCRIPTION:
Persons working in a military unit in Boden and persons connected to the Department of Sports Medicine in Umeå were invited to participate in this study. Only persons older than 18 years was included in the study. The persons included received one bottle of study medicine, a home protocol (WURSS 21) and a viral sampling kit. Whenever the included persons were sure that they had received an episode of common cold they were told to perform a viral sampling from the nose, fill in the protocol and start to use the nasal spray several times daily for one week. The treatment was either a) a saline solution with 5% glucose or b) a saline solution with 200U/ml of glucose oxidase and 5%glucose (active treatment group). The combination of glucose oxidase and glucose produces an acid environment, imitating the effect of the normal nasal flora and Human Rhinoviruses are sensitive to an acid environment. After one week of treatment and daily records of the WURSS 21 protocol the persons returned the spray bottles (Bag-on-Valve), the virus vials and the protocols.

A total of 146 persons were included in the study and 98 persons returned protocols.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Ongoing allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krister Tano, MD,PhD, Principal Investigator — Umeå University
Locations (2):
- Sweden (2):
  - Försvarshälsan, Boden
  - Idrottsmedicin, Umeå

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saline+Glucose Nasal Spray | Nasal Spray With Glucose Oxidase+Glucose
Started | 73 | 73
Completed | 48 | 50
Not Completed | 25 | 23
Not completed — No episode of common cold | 25 | 23

BASELINE CHARACTERISTICS:
Population: Healthy adult volunteers. One part of the included participants was from an education in elite skiing at the University and one part was from a military unit. The participants were told to start the treatment as soon as they were convinced that they had caught a common cold
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline+Glucose Nasal Spray | Nasal Spray With Glucose Oxidase+Glucose | Total
Number analyzed (Participants) | 48 | 50 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 48 | 95
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] | 38 [19 to 72] | 40 [18 to 70] | 39 [18 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 28 | 58
  Male | 18 | 22 | 40
Region of Enrollment [Number; unit: participants]
  Sweden | 48 | 50 | 98

OUTCOME MEASURES:

1. Primary Outcome: Reducing Symptoms of a Common Cold
Description: Using the Wisconsin Upper Respiratory Symptom Score (WURSS-21)it is possible to assess if a nasal spray containing glucose oxidase and glucose would be able to reduce symptoms of a common Cold.
  WURSS 21 is a validated tool of calculating the degree of common Cold symptoms. It consists of 21 questions (20 questions are possible to evaluate) which are graded from 0 to 7 (worst degree of symptoms). These 20 questions (sum of all symptoms) are evaluated every day, Min value is thus 0 and max value/person/day is 140. It is thus possible to calculate the mean value of sum of symptoms for each day in the both groups.
Time Frame: One week
Population: Only the participants that fullfilled the study and who had a positive virus sample (Influensa and adenoviruses excluded) were included in the results. These are the participants that are supposed to benefit from a nasal spray with GO.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Saline+Glucose Nasal Spray | Nasal Spray With Glucose Oxidase+Glucose
Number analyzed (Participants) | 17 | 13
units on a scale
  Start value | 53 [22 to 84] | 53 [23 to 77]
  Value day 1 | 55 [22 to 85] | 54 [30 to 88]
  Value day 2 | 55 [23 to 84] | 49 [28 to 86]
  Value day 3 | 40 [6 to 85] | 36 [7 to 66]
  Value day 4 | 31 [0 to 77] | 29 [1 to 48]
  Value day 5 | 22 [0 to 73] | 20 [0 to 51]
  Value day 6 | 14 [0 to 59] | 14 [0 to 58]
  Value day 7 | 10 [0 to 56] | 12 [0 to 58]

ADVERSE EVENTS:
Time Frame: January 2013 to May 2013
Arm/Group | Saline+Glucose Nasal Spray | Nasal Spray With Glucose Oxidase+Glucose
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/50
Other Adverse Events (participants affected / at risk) | 0/48 | 0/50

LIMITATIONS AND CAVEATS:
Too few virus positive persons in order to get significant results. Local side effects were mild and about the same as in the placebo Group. Influensa season and few rhinovirus infections.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No